CLINICAL TRIAL: NCT04145687
Title: Metformin In Prevention Of Lupus Nephritis In High Risk Patients
Brief Title: Metformin In Prevention of Lupus Nephritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Ting Li, Prof., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Met LN
Record Dates: First submitted 2019-10-22; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500mg tid

SUMMARY:
Lupus nephritis (LN) is a main manifestation of systemic lupus erythematosus (SLE), which will largely effect the prognosis of SLE patients. Our previous 10-year data showed that the development of LN is most common in the first year of SLE, occupying about 17%. And our group has established a prediction model to predict the 1-year probability of LN for SLE patients without renal involvement. Our previous proof-of-concept trial and multicenter, randomized, double-blind, placebo-controlled trial indicated that metformin seemed to have potential to reduce the new-onset of LN in SLE patients (Unpublished data, in review). So the investigators tried to illustrate whether metformin has effect to prevent the development of lupus nephritis in high risk SLE patients based on LN prediction model.

ELIGIBILITY:
Inclusion Criteria:

* New-onset of SLE (within 1 year)
* Meet the 1997 ACR criteria of SLE
* 1-year risk of developing LN higher than 50% based on LN prediction model.
* All the patients received standard care of therapy. (mycophenolate/azathioprine/cyclosporin/tacrolimus/methotrexate/leflunomide were allowed).
* Sign the informed consent.

Exclusion Criteria:

* Patients with kidney involvement at screening were excluded
* Patients with severe SLE were excluded, such as neuropsychiatric and cardiac involvement
* Cyclophosphamide or biologics were not allowed.
* Alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 2 times upper normal limits; creatinine clearance rate < 60ml/min;
* Previous exposure of metformin within 30 days before screening; or previous history of intolerant to metformin;
* Patients who diagnosed of diabetes mellitus;
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Prevention of new-onset LN | 12 months
  Percentage of patients with new-onset lupus nephritis

SECONDARY OUTCOMES:
Change of SLEDAI score | 12 months
  Change of SLEDAI score during follow-up
Change of Prednisone | 12 months
  Change of Prednisone during follow-up
Time to onset of LN | 12 months
  Time to new-onset of lupus nephritis
Change of proteinuria | 12 months
  Change of 24-hour proteinuria during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fangfang Sun, MD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No